CLINICAL TRIAL: NCT01106703
Title: The Effects of PG102 on Allergy-related Risk Factors: A Randomized, Double Blind, Placebo Controlled Study
Brief Title: The Effects of PG102, a Water Soluble Extract From Actinidia Arguta, on Serum Total IgE Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A060655
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Asymptomatic Subjects With Atopy and Elevated Serum IgE
Keywords: atopy, IgE
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG102 group (Experimental)
  Interventions: Dietary Supplement: PG102, a water soluble extract from Actinidia arguta
- placebo group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: PG102, a water soluble extract from Actinidia arguta — PG102 two tables(Actinidia arguta extract:Microcrystalline cellulose(1:1)mixed powder 1120mg) twice a day for 8weeks
  Arms: PG102 group
Other: placebo — placebo two tables(equivalent dose of Microcrystalline cellulose) twice a day for 8weeks
  Arms: placebo group

SUMMARY:
The aim of this study was to evaluate the efficacy of PG102 at lowering levels of total IgE in asymptomatic subjects with atopy.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have atopy but no allergy-related symptoms
* subjects with total IgE levels of 300IU/ml or more
* acquisition of written informed consent prior to commencement of study
* no serious clinical symptoms and normal laboratory test results; in case of abnormal finding, subjects whose conditions are not deemed severe from the judgement of investigators

Exclusion Criteria:

* individuals with normal levels of total serum IgE
* ue of one or more allergic drugs
* serious clinical conditions (such as malignancies, severe cardiovascular disease etc.)
* serious mental disorder
* pregnant woman or woman of childbearing potential within 3 months
* subjects who participated in other clinical trials in the past 6months
* individuals who have a plan to participate in another clinical trials during this trial
* subjects with a history of kiwi allergy
* subjects whose conditions are inappropriate by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
serum total IgE level | 8weeks

SECONDARY OUTCOMES:
serum level of allergy-related factors, such as eosinophilic cation protein(ECP), eotaxin, thymus, and activation-regulated chemokine (TARC), IL-4, IL-5, and IL-13, skin test(atopy score), and adverse reactions | 8weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Up Min, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Soeul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul